CLINICAL TRIAL: NCT06343779
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Cross-over Study of Oral Deucrictibant Soft Capsule for On-Demand Treatment of Attacks in Adolescents and Adults With Hereditary Angioedema
Brief Title: Study of Oral Deucrictibant Soft Capsule for On-Demand Treatment of Angioedema Attacks in Adolescents and Adults With Hereditary Angioedema
Acronym: RAPIDe-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharvaris Netherlands B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHA022121-C306
Record Dates: First submitted 2024-03-18; First posted 2024-04-03 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Hereditary Angioedema; Hereditary Angioedema Type I; Hereditary Angioedema Type II; Hereditary Angioedema Types I and II; Hereditary Angioedema Attack; Hereditary Angioedema With C1 Esterase Inhibitor Deficiency; Hereditary Angioedema - Type 1; Hereditary Angioedema - Type 2; C1 Esterase Inhibitor [C1-INH] Deficiency; C1 Esterase Inhibitor Deficiency; C1 Esterase Inhibitor, Deficiency of; C1 Inhibitor Deficiency; Hereditary Angioedema - Type 3; Hereditary Angioedema Type III
Keywords: HAE; HAE Type I; HAE Type II; Oral Treatment; Bradykinin B2 Receptor Antagonists; PHVS416; PHA121; On-Demand; Deucrictibant; Pharvaris; HAE Type III
MeSH Terms: conditions — Angioedemas, Hereditary; Hereditary Angioedema Types I and II; Hereditary Angioedema Type III

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Deucrictibant administered for first HAE attack, placebo administered for second HAE attack.
  Interventions: Drug: Deucrictibant, Placebo
- Arm 2 (Experimental): Placebo administered for first HAE attack, deucrictibant administered for second HAE attack.
  Interventions: Drug: Deucrictibant, Placebo

INTERVENTIONS:
Drug: Deucrictibant, Placebo — Deucrictibant Soft Capsules for Oral Use

SUMMARY:
This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled, 2-period, 2-treatment cross-over study to evaluate the efficacy and safety of orally administered deucrictibant compared to placebo for the on-demand treatment of HAE attacks, including non-severe laryngeal attacks, in participants ≥12 to ≤75 years of age with HAE type 1, type 2, or type 3, a proportion of whom are using long-term prophylactic medication for HAE.

DETAILED DESCRIPTION:
The study consists of a Screening Phase during which eligibility is confirmed, a Treatment Phase in which participants will be randomized and receive double blinded study drug to treat 2 qualifying HAE attacks (i.e., 2 Treatment Periods within the Treatment Phase), and an End-of-Study Follow-up Phase after the second attack treated with study drug. In addition, for adolescent participants (age ≥12 to <18 years), PK samples are collected after administration of deucrictibant at Day 1 in a non-attack state.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent/assent.
2. Male or female, aged ≥12 to ≤75 years at the time of providing written informed consent/assent.
3. Diagnosis of HAE-1/2/3.
4. History of at least 2 HAE attacks in the last 3 months before screening.
5. Experience with using standard-of-care treatment to effectively manage on-demand treatment for HAE attacks.
6. Participants on long-term prophylactic therapy with plasma-derived C1-INH (danazol, anti-fibrinolytics, berotralstat, or lanadelumab) must be on a stable dose and regimen and intend to remain on the same dose for 6 months before screening and the duration of the study. OR, Participant has stopped using plasma-derived C1-INH (danazol, anti-fibrinolytics, berotralstat) at least 2 weeks or lanadelumab at least 10 weeks before screening.
7. Capable of recording, without assistance, electronic HAE diary and ePRO data using an electronic device.
8. For adolescent participants aged ≥12 and <18 years of age: body weight ≥40 kg.
9. Female participants of childbearing potential must agree to the protocol specified pregnancy testing and contraception methods.

Exclusion Criteria:

1. Any female who is pregnant, plans to become pregnant, or is breastfeeding.
2. Any diagnosis of angioedema other than HAE.
3. Any clinically significant comorbidity or systemic dysfunction that would interfere with the participant's safety or ability to participate in the study.
4. Use of attenuated androgens for short-term prophylaxis within 2 weeks before screening.
5. Abnormal hepatic function.
6. Abnormal renal function (eGFR <60 ml/min/1.73 m2).
7. History of alcohol or drug abuse within the previous year, or current evidence of substance dependence or abuse.
8. Has received prior on-demand HAE treatment with deucrictibant.
9. Currently participating in any other investigational drug study or receiving other investigational treatment within the last 30 days, or within 5 half-lives (whichever is longer) of the time of randomization.
10. Prior gene therapy for any indication at any time.
11. Use of concomitant medications with systemic absorption that are strong inhibitors of CYP3A4 or strong inducers of CYP3A4 within the last 30 days, or within 5 half-lives (whichever is longer) of the time of randomization.
12. Known hypersensitivity to study drug or any of the excipients of study drug.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
Time to onset of symptom relief, defined as Patient Global Impression of Change (PGI-C) rating of at least "a little better" for 2 consecutive timepoints within 12 hours post-treatment. | Pre-treatment to 12 hours post-treatment.
  The PGI-C (7-point scale) is used to evaluate the change in the HAE attack symptoms as compared to pre-treatment.

SECONDARY OUTCOMES:
Proportion of study drug-treated attacks achieving PGI-C rating of at least "a little better" at 4 hours post-treatment. | Pre-treatment to 4 hours post-treatment.
  The PGI-C (7-point scale) is used to evaluate the change in the HAE attack symptoms as compared to pre-treatment.
Time to substantial symptom relief, defined as achieving PGI-C rating of at least "better" for 2 consecutive timepoints within 12 hours post-treatment. | Pre-treatment to 12 hours post-treatment.
  The PGI-C (7-point scale) is used to evaluate the change in the HAE attack symptoms as compared to pre-treatment.
Time to substantial symptom relief by Patient Global Impression of Severity (PGI-S). | Pre-treatment to 12 hours post-treatment.
  Defined as achieving ≥1 point reduction in PGI-S (5-point scale) from pre-treatment for 2 consecutive timepoints within 12 hours post-treatment.
Time to complete symptom resolution, defined as achieving PGI-S rating of "none" within 48 hours post-treatment. | Pre-treatment to 48 hours post-treatment.
  The PGI-S (5-point scale) is used to evaluate the severity of HAE attack symptoms.
Time to End of Progression (EoP) in attack symptoms within 12 hours. | Pre-treatment to 12 hours post-treatment.
  EoP time defined as the earliest post-treatment timepoint after which all subsequent PGI-C ratings are stable or improved.
Proportion of study drug-treated attacks requiring rescue medication within 24 hours post-treatment. | Pre-treatment to 24 hours post-treatment.
  Rescue medication is defined as the participant's usual acute on-demand HAE treatment taken if symptoms persist or progress after study drug administration.
Proportion of attacks achieving symptom resolution. | Pre-treatment to 24 hours post-treatment.
  Defined as achieving PGI-S rating of "none" with one dose of study drug at 24 hours post-treatment.
Time to substantial symptom relief by Angioedema Symptom Rating Scale (AMRA). | Pre-treatment to 12 hours post-treatment.
  Defined as a ≥50% reduction in AMRA composite score from pre-treatment for 2 consecutive timepoints within 12 hours post-treatment.
Time to almost complete or complete symptom relief by AMRA. | Pre-treatment to 24 hours post-treatment.
  Defined as all item scores in AMRA having a value ≤10 for 2 consecutive timepoints within 24 hours post-treatment.
Proportion of study drug-treated attacks reaching almost complete or complete symptom relief by AMRA. | Pre-treatment to 24 hours post-treatment.
  Defined as all item scores in AMRA having a value ≤10 at 24 hours post-treatment.
Time to EoP in attack symptoms within 12 hours. | Pre-treatment to 12 hours post-treatment.
  Defined as the earliest post-treatment timepoint after which every individual AMRA item is stable or improved at all subsequent timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Pharvaris, Study Director — Pharvaris Netherlands B.V.
Locations (69):
- United States (13):
  - Study Site, Birmingham, Alabama
  - Study Site, Paradise Valley, Arizona
  - Study Site, Little Rock, Arkansas
  - Study Site, San Diego, California
  - Study Site, Santa Monica, California
  - Study Site, Walnut Creek, California
  - Study Site, Colorado Springs, Colorado
  - Study Site, Chevy Chase, Maryland
  - Study Site, Boston, Massachusetts
  - Study Site, Detroit, Michigan
  - Study Site, St Louis, Missouri
  - Study Site, Hershey, Pennsylvania
  - Study Site, Dallas, Texas
- Argentina (2):
  - Study Site, Buenos Aires
  - Study Site, Salta
- Australia (2):
  - Study Site, Campbelltown, New South Wales
  - Study Site, Box Hill
- Austria (3):
  - Study Site, Graz
  - Study Site, Linz
  - Study Site, Vienna
- Brazil (5):
  - Study Site, Paraná
  - Study Site, Ribeirão Preto
  - Study Site, Salvador
  - Study Site, Santo André
  - Study Site, São Paulo
- Study Site, Sofia, Bulgaria
- Study Site, Edmonton, Alberta, Canada
- Colombia (2):
  - Study Site, Bogotá
  - Study Site, Medellín
- Study Site, Brno, Czechia
- France (2):
  - Study Site, Lille
  - Study Site, Paris
- Germany (3):
  - Study Site, Berlin
  - Study Site, Frankfurt am Main
  - Study Site, Lübeck
- Study Site, Hong Kong, Hong Kong
- Study Site, Budapest, Hungary
- Study Site, Dublin, Ireland
- Italy (5):
  - Study Site, Catania
  - Study Site, Milan
  - Study Site, Padua
  - Study Site, Palermo
  - Study Site, Roma
- Japan (5):
  - Study Site, Chiba
  - Study Site, Hiroshima
  - Study Site, Kanagawa
  - Study Site, Osaka
  - Study Site, Tokyo
- Study Site, Amsterdam, Netherlands
- Study Site, Skopje, North Macedonia
- Study Site, Krakow, Poland
- Study Site, San Juan, Puerto Rico
- Study Site, Sângeorgiu de Mureş, Romania
- Study Site, Riyadh, Saudi Arabia
- Study Site, Singapore, Singapore
- Study Site, Cape Town, South Africa
- South Korea (2):
  - Study Site, Daegu
  - Study Site, Seoul
- Study Site, Barcelona, Spain
- Study Site, Lund, Sweden
- Turkey (Türkiye) (3):
  - Study Site, Ankara
  - Study Site, Istanbul
  - Study Site, Izmir
- United Kingdom (6):
  - Study Site, Bristol
  - Study Site, Camberley
  - Study Site, Cambridge
  - Study Site, Leeds
  - Study Site, London
  - Study Site, Plymouth